CLINICAL TRIAL: NCT05686824
Title: Exploring the Attrition and Retention of Midwifery Professionals and Identifying Lessons for the Future: an Organisational Case Study
Brief Title: Midwifery Retention Project
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: NHS Devon ICB (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRAS 321453
Record Dates: First submitted 2023-01-06; First posted 2023-01-17 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Retention/Attrition of Midwives
Keywords: retention, attrition, midwifery, workforce, NHS
MeSH Terms: conditions — Tooth Wear; Nance-Horan syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Midwives and student midwives at one Trust: No intervention - this is an exploratory case study

SUMMARY:
The NHS is experiencing a significant workforce crisis across the service; with currently >130, 000 vacancies, therefore, national efforts to improve recruitment and retention are a priority. In maternity services, there are currently 2,500 WTE midwife vacancies and over three-quarters of Heads of Midwifery cite it is 'increasingly difficult' to fill these vacancies . A vital component of a sustainable workforce and safe maternity care is retaining newly qualified midwives (where attrition is currently high) and experienced midwives already working within the service. However, data repeatedly demonstrate dissatisfaction and intentions to leave the midwifery profession. Recognising the importance of retention, NSHEI allocated a one-off lump sum of £50,000 to each hospital Trust to specifically employ midwives to support retention efforts. However, to date, research has not captured contemporary midwifery attrition and retention insights with this role in place. Therefore, the purpose of this study is to capture, analyse and disseminate localised data from one NHS Trust to inform future local, regional and national retention projects. Specifically, this study aims to explore the views of midwives and student midwives at Torbay and South Devon NHS Foundation Trust regarding intentions to stay or leave either their current workplace and/or the profession. These subtle but salient differences are important as some may prefer to work elsewhere but remain in midwifery, conversely, others may be satisfied with their workplace but intend to leave the profession. We will also gather insights regarding the retention midwife role, their work to date and potential impact. We will gather the data via documentary review, a survey aimed at midwives and student midwives and 10-15 individual interviews. Using these insights, we will identify recommendations for the local, regional and national workstreams to inform future retention work.

DETAILED DESCRIPTION:
The broad purpose of this study is to generate insights regarding the attrition and retention of midwives within a specific organisation (Torbay and South Devon NHS Trust) to inform future staffing retention quality improvement projects, locally and nationally.

A single case study approach is the chosen methodology for this research. This is an appropriate approach as it seeks to 'investigate contemporary phenomena within its real-life context' and to generate in-depth and multi-faceted understandings (explaining, describing or exploring) of complex issues within a naturalistic context; which in this study, relates to the attrition and retention of midwives employed by a specific Trust. While these issues are not unique to this Trust, therefore, is not an intrinsic case study, their willingness to explore these issues means an 'instrumental' case study will facilitate 'a broader appreciation of [the] issue or phenomenon'.

This case study is focused on midwifery retention and recruitment, as such, eligible participants will be all midwives currently employed within the Trust. For those on maternity or sick leave but wish to participate, they too will be eligible. Additionally, we will include student midwives currently placed within Torbay and South Devon NHS Foundation Trust. All student midwives will be eligible to participate in the survey but only 3rd year midwives will be eligible for an interview.

Recruitment will consist of purposive and snowball methods via the retention midwife leads, internal social media, internal work emails and adverts placed within the Trust. Adverts will include information about the interview option (midwives and 3rd year student midwives only) and the survey which will include a link and/or QR code to the survey for instant access (all midwives and student midwives eligible).

Informed consent for the survey will be obtained via the first page of the Qualtrics survey whereby all appropriate information regarding the study and how the data will be stored and used will be stated. Participants will be able to opt in to complete the survey or opt out by simply closing the survey. Participants will be advised they will not be able to withdraw from the study after submitting their responses as the data is anonymised, we will not be able to accurately delete their information.

Informed consent for the online interview will be obtained at the start of the meeting, prior to any demographic or interview questions. It is expected that the participant information sheet will have been read prior to the interview as this will be sent out during an initial inquiry contact. At the start of the interview, the researchers will check whether the participants have questions or queries that need to be clarified. The consent form will be carried out 'virtually' together, with the researcher sharing the screen, asking each question and signing on behalf of the participant, and this will be recorded. Participants will be advised that they can stop the interview at any time and have the right to withdraw their data within two weeks of the interview (prior to analysis starting).

We don't foresee particular risks to this research, although we have considered:

Ethical considerations during recruitment relates to maintaining confidentiality for some participants may not wish to disclose their participation to their wider teams. Therefore, to mitigate against this, the recruitment emails and adverts will include, either a direct link/QR code the survey and the researchers direct contact details to arrange interviews. This way, no one outside of the research team will be aware of who has participated, nor will this information be disclosed.

Ethical considerations during the interview relate to two possibilities: a) if a participant becomes distressed during the interview, the researcher will offer to stop the interview immediately and offer a referral to their Professional Midwifery Advocate; b) should the participant, a registered health professional, reveal dangerous or illegal practice, the interview will be stopped, and they will be advised a referral to their senior leaders made. The latter possibility is highly unlikely.

Survey confidentiality will be maintained as it will be anonymous. Interview recordings, once downloaded will have a pseudonym applied and the recording deleted. Following transcription, the manuscripts any identifying features (names, places, personal details) will be removed prior to analysis.

ELIGIBILITY:
Inclusion Criteria:

* employed midwives at Torbay Hospital.
* student midwives on placement at Torbay Hospital.

Exclusion Criteria:

* Midwives or student midwives not working/placed at Torbay Hospital.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Midwives and student midwives
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Survey | 2 weeks
  To explore midwives and student midwives views on leaving or staying within their workplace and/or the profession.
Interview | 6 weeks
  Follow up questions to explore midwives intentions to leave or stay within their hospital Trust and/or profession.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Feeley, PhD, Principal Investigator — King's College London
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No